CLINICAL TRIAL: NCT04158713
Title: Chemoprevention With Monthly IPTp With Dihydroartemisinin-piperaquine for Malaria in HIV-infected Pregnant Participants on Daily Cotrimoxazole in Kenya and Malawi: a Multi-centre Placebo-controlled Trial
Brief Title: Improving PRegnancy Outcomes With PReVEntive Therapy in Africa-2 (IMPROVE-2)
Acronym: IMPROVE-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Kenya Medical Research Institute (Other); Kamuzu University of Health Sciences (Other); Kenya National AIDS & STI Control Programme (Other); KEMRI-Wellcome Trust Collaborative Research Program (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); University of Copenhagen (Other); University of Cape Town (Other); University of Massachusetts, Worcester (Other); University of Toronto (Other); University of Melbourne (Other); CardiaBase (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 17-005
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Pregnancy; HIV; Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: Allocation: randomised; intervention model: parallel assignment; arms: 2; allocation ratio: 1:1; stratified by site (hospital) and HIV-status (known-positive and newly-diagnosed). Masking: Placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTX-alone (Placebo Comparator): Daily, one double-strength tablet of 160mg of sulfamethoxazole and 800mg of trimethoprim plus monthly placebo-DP, given as a fixed dose of 3 placebo-DP tablets daily for three days until delivery.
  Interventions: Drug: Intermittent Preventive Therapy with Dihydroartemisinin-Piperaquine
- CTX-DP (Experimental): Daily, one double-strength tablet of 160mg of sulfamethoxazole and 800mg of trimethoprim plus monthly DP, given as a fixed dose of 3 tablets (40 mg of dihydroartemisinin and 320 mg of piperaquine) daily for three days until delivery.
  Interventions: Drug: Intermittent Preventive Therapy with Dihydroartemisinin-Piperaquine

INTERVENTIONS:
Drug: Intermittent Preventive Therapy with Dihydroartemisinin-Piperaquine — Monthly DP fixed dose of 3 tablets (40 mg of dihydroartemisinin and 320 mg of piperaquine) daily for three days until delivery. All participants will (continue to) receive daily cotrimoxazole (CTX) (one double-strength tablet of 160mg of sulfamethoxazole and 800mg of trimethoprim) and anti-retroviral drugs.
  Other Names: Monthly DP; D-artepp

SUMMARY:
2.3.3 Short technical protocol summary Background: Pregnant women represent a vulnerable population for malaria. HIV-infected women are particularly at risk. In HIV-infected pregnant women, WHO recommends daily cotrimoxazole (CTX), an antifolate drug, for malaria chemoprevention and prophylaxis against opportunistic infection. However, there is cross-resistance with sulphadoxine-pyrimethamine (SP), and high levels of antifolate resistance threatens the antimalarial effect of CTX. Recent trials with intermittent preventive therapy (IPT) with mefloquine in HIV-infected women on daily CTX, suggested that chemoprevention with an effective antimalarial markedly improves the protection against malaria compared to daily CTX alone. However, mefloquine was not well tolerated.

The long-acting combination of dihydroartemisinin-piperaquine (DP) is well tolerated and has shown great promise as IPTp in HIV-negative women in East-Africa. Chemoprevention with monthly DP has also been explored in HIV-infected pregnant women on daily CTX in Uganda. Unfortunately, the study was inconclusive because malaria transmission was too low and a clinically relevant drug interaction with efavirenz (EFV) was found reducing the exposure to DP. WHO now recommends dolutegravir (DTG) based combination antiretroviral therapy (ARTs) as the preferred firstline regimen including for pregnant women in the 2nd and 3rd trimester of pregnancy for the prevention of mother-to-child transmission of HIV. As a result, many countries in Africa are now transitioning to DTG-based combination antiretroviral therapy (cARTs). No such drug-drug interaction is expected between DTG and DP. We will, therefore, assess the safety and efficacy of malaria chemoprevention with monthly DP in HIV-infected women on daily CTX and DTG-based cARTs.

Objectives and methods: This is a 2-arm, individually-randomized, multi-centre, placebo-controlled superiority trial comparing the safety and efficacy of daily CTX plus monthly DP ('CTX-DP') versus daily CTX plus monthly placebo-DP (i.e. 'CTX-alone', control arm) to reduce malaria and the adverse effects of malaria in 898 (449 per arm) HIV-infected pregnant women on DTG-based cARTs. The study will be conducted in 8 hospitals in Kenya and Malawi in high SP-resistance areas with a high prevalence of malaria. These are the same sites where the sister trial in HIV-uninfected women is being conducted in Kenya and Malawi (IMPROVE trial). Both the mother and baby will be followed for 6-8 weeks after delivery. The study is powered at 80% (alpha=0.05) to detect ≥50% relative risk reduction (RR=0.50) in the primary outcome (cumulative incidence of malaria infection) from 12% in the CTX-alone arm (control arm) to 6% in in the interventions arm allowing for 20% non-contributors. The trial includes a pharmacokinetic assessment, cardiac monitoring for safety, assessment of antimalarial drug and the impact on immune responses to malaria and other pathogens.

DETAILED DESCRIPTION:
2.3.4 Long technical protocol summary Title: Chemoprevention with monthly IPTp with dihydroartemisinin-piperaquine for malaria in HIV-infected pregnant participants on daily cotrimoxazole in Kenya and Malawi: a multi-centre placebo-controlled trial(IMPROVE-2).

Background and rationale: In malaria-endemic Africa, HIV and malaria conspire to increase the risks of adverse pregnancy outcomes. For HIV-infected pregnant women, WHO recommends daily cotrimoxazole (CTX) for chemoprevention for malaria and prophylaxis against opportunistic infection. However, there is cross-resistance with SP, and high levels of antifolate resistance threaten the antimalarial effect of CTX. Recent trials in HIV-infected pregnant women who received daily CTX plus IPTp with mefloquine, suggested that chemoprevention with an effective antimalarial markedly reduces the risk of malaria compared to daily CTX alone. However, mefloquine was not well tolerated. The long-acting combination of dihydroartemisinin-piperaquine (DP) is well tolerated and has shown great promise as IPTp in HIV-negative women in East-Africa. Chemoprevention with monthly DP has also been explored in HIV-infected women on daily CTX in Uganda. Unfortunately, the study was inconclusive as malaria transmission was too low. Furthermore, a clinically relevant drug-drug interaction between DP and efavirenz (EFV) was found to reduce DP drug levels. Following the recommendation from WHO, many countries in Africa are transitioning from EFV-based to dolutegravir (DTG) based combination antiretroviral therapy (cARTs). WHO now recommends DTG-based cARTS as the preferred first-line cART regimen in the 2nd and 3rd trimester of pregnancy. No such drug-drug interaction is expected between DTG and DP. We will therefore assess the safety and efficacy of malaria chemoprevention with monthly DP in HIV-infected women on daily CTX and DTG-based cARTs. We will therefore assess the safety and efficacy of malaria chemoprevention with monthly IPTp with DP in women on daily CTX and DTG-based cARTs and daily CTX.

Overall aim: To provide WHO with evidence on whether monthly IPTp-DP can improve current policies to control malaria in HIV-infected pregnant women on daily CTX in areas with high levels of parasite resistance and malaria in East and Southern Africa.

Primary objective: To determine if monthly IPTp-DP in HIV-infected pregnant women receiving daily CTX is safe and superior to daily CTX-alone for controlling malaria infection in areas with high antifolates resistance to SP and CTX in Malawi and Kenya.

Hypotheses: Monthly IPTp-DP in women receiving daily CTX is superior to daily CTX-alone in controlling malaria infection during pregnancy in HIV infected women on antiretroviral therapy.

Overview Study Design: This multi-centre trial will be conducted in antenatal clinics in 8 hospitals in Kenya and Malawi located in areas with high prevalence of HIV and malaria and with high anti-folate resistance of the malaria parasite. These are the same sites where the sister trial in HIV-uninfected women (all gravidae) is being conducted in Kenya and Malawi (IMPROVE trial: NCT03208179). Overall, 898 (449 per arm) HIV-infected pregnant women who are 16 to 28 weeks pregnant assessed by ultrasound dating, will be randomised to receive one of the two interventions. Permuted block randomisation stratified by site (i.e. hospital) and HIV-status (known-positive and newly-diagnosed) will be used. Allocation concealment will be ensured by using sequentially numbered, sealed, opaque envelopes. The study will include pharmacokinetic studies and cardiac monitoring in a sub group of women. Other components include molecular marker studies of antimalarial resistance. We will also look at the impact on biomarkers of placental function and trans-placental antibody transfer and multi-pathogen neonatal cell mediated immune responses.

Study Interventions: Daily CTX for all trial participants receiving cARTs in addition to: a) monthly-DP ('CTX-DP'), or b) monthly DP-placebo ('CTX-alone') (control).

Follow-up procedures: Monthly visits during pregnancy, and then at delivery. Mother and newborn follow-up at 7 days and 6-8 weeks post-partum.

Primary outcome: The cumulative incidence of malaria infection detected from 2 weeks after the first day of the first dose of the first course to delivery inclusive, defined as the presence of peripheral (maternal) or placental (maternal) Plasmodium infection detected by either molecular diagnostics (henceforth referred to as PCR), microscopy, RDT or placental histology (active infection).

Sample size: 898 (449 per arm), allowing for 20% loss to follow-up. Data Analysis: Log-binomial regression will be used to analyse the primary outcome, controlled for site and gravidity.

Primary partner institutions: KEMRI, Kenya; College of Medicine, University of Malawi, Malawi; Liverpool School of Tropical Medicine (LSTM); London School of Hygiene and Tropical Medicine (LSHTM); US Centers for Disease Control and Prevention (CDC); University of Bergen, Norway.

Funding: Joint Global Health Trials Scheme, Medical Research Council/Wellcome Trust/DFID, UK; and the European and Developing Countries Clinical Trials Partnership (EDCTP).

Sponsor: Liverpool School of Tropical Medicine (LSTM); Pembroke Place, Liverpool L3 5QA, UK, Phone: +44 0151 7053794; Email: lstmgov@lstmed.ac.uk.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected pregnant women between 16-28 weeks' gestation
* Viable singleton pregnancy
* On or eligible for cARTs and CTX
* A resident of the study area
* Willing to adhere to scheduled and unscheduled study visit procedures
* Willing to deliver in a study clinic or hospital
* Provide written informed consent

Exclusion Criteria:

* Multiple pregnancies (i.e. twin/triplets)
* HIV-negative or HIV status unknown
* Known heart ailment
* Severe malformations or non-viable pregnancy if observed by ultrasound
* Participants with advanced HIV-disease at WHO clinical stage 3 and 4
* Confirmed or suspected TB infection,
* Unable to give consent
* Known allergy or contraindication to any of the study drugs

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 898 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of malaria infection | Detected from 2 weeks after the first day of the first dose of the first course to delivery inclusive. The total duration of the trial is 24 months. Actual participant recruitment and follow up is expected to take up to 19 months.
  The primary outcome will be the cumulative incidence of malaria infection detected from 2 weeks after the first day of the first dose of the first course to delivery inclusive, defined as the presence of peripheral (maternal) or placental (maternal) Plasmodium infection detected by either molecular diagnostics (henceforth referred to as PCR), microscopy, RDT or placental histology (active infection).

SECONDARY OUTCOMES:
Efficacy of the intervention on the following listed secondary outcomes | The total duration of the trial is 24 months. Actual participant recruitment and follow up is expected to take up to 19 months (12 months recruitment plus 7 months of mother-infant follow-up until the child is 6 weeks old
  1. Incidence of malaria infection
  2. The individual components of the composite malaria infection endpoints
  3. Incidence of clinical malaria.
  4. Malaria infection at delivery
  5. Placental malaria by histology (active, past, and active and past infections pooled)
  6. Placental malaria by any measure
  7. Maternal peripheral malaria infection at delivery by any measure
  8. Placental inflammation or chorioamnionitis
  9. Adverse pregnancy outcome: the composite of foetal loss (spontaneous abortion or stillbirth), or singleton live births born small-for-gestational-age (SGA), or with low birthweight (LBW), or preterm (PT) (SGA-LBW-PT), or subsequent neonatal death by day 28.
  10. Composite of foetal loss and neonatal mortality.
  11. SGA-LBW-PT composite.
  12. The individual components of the above composites
  13. Neonatal length and stunting.
  14. Evidence of arboviral infections
Safety: Cardiac safety, serious adverse events and MTCT of HIV | The total duration of the trial is 24 months. Actual participant recruitment and follow up is expected to take up to 19 months (12 months recruitment plus 7 months of mother-infant follow-up until the child is 6 weeks old
  1. QTc-prolongation.
  2. Congenital malformations.
  3. Maternal mortality
  4. Other SAEs and AEs.
  5. Mother to child transmission of HIV
Tolerance | The total duration of the trial is 24 months. Actual participant recruitment and follow up is expected to take up to 19 months (12 months recruitment plus 7 months of mother-infant follow-up until the child is 6 weeks old
  1. History of vomiting study drug (<30 min).
  2. Dizziness.
  3. Gastrointestinal complaints.
Antimicrobial activity and resistance | The total duration of the trial is 24 months. Actual participant recruitment and follow up is expected to take up to 19 months (12 months recruitment plus 7 months of mother-infant follow-up until the child is 6 weeks old
  Frequency of molecular markers of drug resistance in Plasmodium falciparum infections during pregnancy and delivery.
Pharmacokinetic parameters | The total duration of the trial is 24 months. Actual participant recruitment and follow up is expected to take up to 19 months (12 months recruitment plus 7 months of mother-infant follow-up until the child is 6 weeks old
  Standard pharmacokinetic parameters for dolutegravir, piperaquine and CTX.

CONTACTS AND LOCATIONS:
Overall Officials: Feiko terKuile, MD-PhD, Principal Investigator — Liverpool School of Tropical Medicine
Locations (1):
- Kenya Medical Research Institute, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Biological samples and data will be shared using material and data transfer agreements with the collaborating institutions (see 2.2.4 Collaborators, page 9) to minimise the risk of unauthorised analysis beyond the scope of the agreed parameters.
Supporting Information: Study Protocol
Time Frame: Five years
Access Criteria: The full protocol will be available on request to any interested professional and may be published in a peer reviewed journal or deposited in an online repository. Individual, de-identified participant data will be made available for meta-analyses as soon as the data analysis is completed, with the understanding that results of the meta-analysis will not be published prior to the results of the individual trial without prior agreement of the investigators. No later than five years after the publication of the trial a fully de-identified data set of the complete patient-level data will be available for sharing purposes, such as via the WWARN repository platform (http://www.wwarn.org/working-together/sharing-data/accessing-data). All requests for data for secondary analysis will be considered by a Data Access Committee to ensure that use of data is within the terms of consent and ethics approval.

REFERENCES:
- [Derived] Pons-Duran C, Wassenaar MJ, Yovo KE, Marin-Carballo C, Briand V, Gonzalez R. Intermittent preventive treatment regimens for malaria in HIV-positive pregnant women. Cochrane Database Syst Rev. 2024 Sep 26;9(9):CD006689. doi: 10.1002/14651858.CD006689.pub3. PMID 39324693
- [Derived] Barsosio HC, Madanitsa M, Ondieki ED, Dodd J, Onyango ED, Otieno K, Wang D, Hill J, Mwapasa V, Phiri KS, Maleta K, Taegtmeyer M, Kariuki S, Schmiegelow C, Gutman JR, Ter Kuile FO. Chemoprevention for malaria with monthly intermittent preventive treatment with dihydroartemisinin-piperaquine in pregnant women living with HIV on daily co-trimoxazole in Kenya and Malawi: a randomised, double-blind, placebo-controlled trial. Lancet. 2024 Jan 27;403(10424):365-378. doi: 10.1016/S0140-6736(23)02631-4. Epub 2024 Jan 12. PMID 38224710

DOCUMENTS (2):
  • Study Protocol (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/13/NCT04158713/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/13/NCT04158713/SAP_001.pdf